CLINICAL TRIAL: NCT01720251
Title: Phase IIb Study to Assess the Efficacy, Safety and Tolerability of Two Dosing Regimens of AllerT in Comparison to Placebo in Adult Subjects Allergic to Birch Pollen
Brief Title: Efficacy Study of a Preseasonal Treatment With AllerT in Subjects With Birch Pollen Allergy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anergis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AN004T; 2011-002259-32 (EudraCT Number)
Record Dates: First submitted 2012-10-29; First posted 2012-11-02 (Estimated); Results first posted 2015-04-13 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-03

CONDITIONS: Allergic Rhinitis; Rhinoconjunctivitis
Keywords: allergic rhinitis; birch pollen; immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- placebo (Placebo Comparator): SC injections of placebo
  Interventions: Drug: placebo
- AllerT low dose (Experimental): SC injections of AllerT 25 or 50 micrograms
  Interventions: Drug: AllerT low dose
- AllerT full dose (Experimental): SC injections of AllerT 50-100 micrograms
  Interventions: Drug: AllerT full dose

INTERVENTIONS:
Drug: placebo — SC injections of placebo on days 1, 7, 14, 28 and 56
  Arms: placebo
Drug: AllerT low dose — SC injections of AllerT 25-50 micrograms on days 1, 7, 14, 28 and 56
  Other Names: AllerT 25-50 micrograms
  Arms: AllerT low dose
Drug: AllerT full dose — SC injections of AllerT 50-100 micrograms on days 1, 7, 14, 28 and 56
  Other Names: AllerT 50-100 micrograms
  Arms: AllerT full dose

SUMMARY:
The main objective of the trial is to demonstrate the efficacy of a two months pre-seasonal treatment with AllerT 100 µg maintenance dose in reducing symptoms of allergic rhinoconjunctivitis during the following birch pollen season

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe allergic rhinoconjunctivitis to birch pollen:

  1. Score of symptoms of the Rhinoconjunctivitis Symptom Score (RSS) ≥ 12 during the two preceding birch pollen seasons
  2. Previous use of anti-allergy medications during the two preceding birch pollen seasons
  3. Positive SPT to birch pollen extract
  4. Positive specific IgE CAP test for Bet v 1

Exclusion Criteria:

* uncontrolled asthma, FEV1 < 80% of predicted
* previous SIT (specific immunotherapy) to birch pollen or any other SIT within 5 years
* clinical symptoms due to allergens other than birch pollen during the whole trial period
* history of anaphylaxis
* positive skin prick test to AllerT
* any other treatment or conditions which may increase the risk of the study for the subject or affect the efficacy assessments during the birch pollen season

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francois Spertini, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (24):
- Denmark (3):
  - Allergiklinikken, Hellerup, Copenhagen
  - Lungemedicinsk Forskningsafdeling, Aarhus
  - Klinisk Institute, Odense
- France (2):
  - CHU de Reims, Reims
  - Hopitaux Universitaires de Strasbourg, Strasbourg
- Latvia (3):
  - Viktorija Vevere private practice of Allergology, Rēzekne
  - Paul Stradins Clinical University Hospital - Pulmonology Allergology, Riga
  - Center of examination and treatment of allergic diseases, Riga
- Lithuania (4):
  - Kaunas Clinics University Hospital, Kaunas
  - Allergy Clinic JSC Perspektyvos, Vilnius
  - Vilnius University Hospital, Vilnius
  - Antakalnio affiliation of the Vilnius City Allergy Center, Vilnius
- Poland (8):
  - SPZOZ Uniwersytecki Szpital Kliniczny - Allergology, Lodz
  - Alergologii Centrum, Lodz
  - Alergotest, Lublin
  - Alergo-Med, Tarnów
  - Centrum Alergologii IRMED, Warsaw
  - Silesian Piasts University of Medicine in Wrocław, Wroclaw
  - Aler-med, Wroclaw
  - NZOZ Przychodnia Lekarska Hipokrates, Zabrze
- Sweden (3):
  - University hospital Skane, Lund
  - Orebro University Hospital, Örebro
  - Lungavdelningen, Vastmanlands, Västerås
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | AllerT Low Dose | AllerT Full Dose
Started | 79 | 79 | 82
Completed | 78 | 77 | 82
Not Completed | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: In AllerT low dose group, one patient has been randomized but not treated explaining the difference beween baseline participants number and participant flow
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AllerT Low Dose | AllerT Full Dose | Total
Number analyzed (Participants) | 79 | 78 | 82 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (9.08) | 36.2 (9.92) | 36.4 (9.36) | 35.6 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 43 | 43 | 124
  Male | 41 | 35 | 39 | 115

OUTCOME MEASURES:

1. Primary Outcome: Combined Rhinoconjunctivitis Symptom and Medication Score
Description: The efficacy analysis will be performed on the symptom and medication data collected from the first day of the birch pollen season as defined by pollen counts in the air in each site region (from March to May 2013 depending on site region), to 42 days later or to the end of the pollen season, whichever comes first.
  The scale range is from 0 to 3. Lower is the the RSMS value, better is the efficacy as this implies that lower is the symptoms and concomitant medication intake by the patient The RSMS includes 2 subscales : the Rhinoconjunctivitis Symptom Score (RSS) with a range of values from 0 to 3 and the Rhinoconjunctivitis Medication Score Score (RMS) with also a range of values from 0 to 3 The RSMS is the sum of the RSS and RMS divided by 2
Time Frame: up to 6 weeks during the birch pollen season 2013
Measure: Mean (Standard Deviation); unit: score (maximum=3)
Arm/Group | Placebo | AllerT Low Dose | AllerT Full Dose
Number analyzed (Participants) | 78 | 77 | 82
score (maximum=3) | 0.86 (0.603) | 0.64 (0.530) | 0.72 (0.573)

2. Secondary Outcome: Quality of Life
Description: mini-RQLQ questionnaires
Time Frame: up to 6 weeks during the birch pollen season 2013
Reporting Status: Not Posted

3. Secondary Outcome: Safety and Tolerability
Description: Adverse events will be collected throughout the trial period and will be reported as Treatment emergent adverse events occurring between start of treatment and 28 days after completion of treatment for each subject
Time Frame: from start of treatment to 28 days after completion of treatment, i.e. for approximately 12 weeks
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Immunological Markers: Specific IgE and IgG4
Description: blood samples will be drawn at the above time points to measure immunological markers: specific IgE and IgG4
Time Frame: before treatment, 4 weeks after the last injection and 2 weeks before, at the peak time and within 2 weeks after the end of the expected birch pollen season 2013
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Placebo: All patients having received at least one injection of Placebo (Safety Set)
- Allert 50 µg: All patients having received at least one injection of Allert 50 µg (Safety Set)
- AllerT 100 µg: All patients having received at least one injection of Allert 100 µg (Safety Set)
Arm/Group | Placebo | Allert 50 µg | AllerT 100 µg
Serious Adverse Events (participants affected / at risk) | 0/79 | 1/78 | 2/82
Other Adverse Events (participants affected / at risk) | 59/79 | 70/78 | 70/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=79) | Allert 50 µg (N=78) | AllerT 100 µg (N=82)
conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Skull fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — considered as non drug-related
Tongue oedema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=79) | Allert 50 µg (N=78) | AllerT 100 µg (N=82)
Injection site pain (Skin and subcutaneous tissue disorders) | 26 | 20 | 16
Injection site reaction (Skin and subcutaneous tissue disorders) | 10 | 19 | 15
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 14 | 13 | 16
Injection site erythema (Skin and subcutaneous tissue disorders) | 18 | 7 | 11
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 7 | 22 | 25
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 17 | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 12 | 26
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 20 | 11
Conjunctivitis (Eye disorders) | 5 | 11 | 12
Injection site oedema (Skin and subcutaneous tissue disorders) | 9 | 8 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI of the trial owns options in the sponsor company and is member of the Board of Anergis SA